CLINICAL TRIAL: NCT06024239
Title: A Multiple Dose Escalation Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of ABBV-932 in Healthy Adult Subjects, Subjects With Generalized Anxiety Disorder (GAD) and Subjects With Bipolar Disorder
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of ABBV-932 in Healthy Adult Participants, Participants With Generalized Anxiety Disorder (GAD) and Participants With Bipolar Disorder (BPD)
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-893
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers; Generalized Anxiety Disorder (GAD); Bipolar Disorder (BPD)
Keywords: ABBV-932; Generalized Anxiety Disorder (GAD); Bipolar Disorder (BPD)
MeSH Terms: conditions — Generalized Anxiety Disorder; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part A, ABBV-932 (Experimental): Participants will receive ABBV-932 once daily (QD) for 14 days.
  Interventions: Drug: ABBV-932
- Part A, Placebo for ABBV-932 (Experimental): Participants will receive placebo for ABBV-932 QD for 14 days.
  Interventions: Drug: Placebo for ABBV-932
- Part B, ABBV-932 (Experimental): Participants will receive ABBV-932 QD for 28 days.
  Interventions: Drug: ABBV-932
- Part B, Placebo for ABBV-932 (Experimental): Participants will receive placebo for ABBV-932 QD for 28 days.
  Interventions: Drug: Placebo for ABBV-932
- Part C, ABBV-932 (Experimental): Participants will receive ABBV-932 QD for 28 days.
  Interventions: Drug: ABBV-932
- Part C, Placebo for ABBV-932 (Experimental): Participants will receive placebo for ABBV-932 QD for 28 days.
  Interventions: Drug: Placebo for ABBV-932
- Part D, ABBV-932 (Experimental): Participants will receive ABBV-932 QD for 42 days.
  Interventions: Drug: ABBV-932
- Part D, Placebo for ABBV-932 (Experimental): Participants will receive placebo for ABBV-932 QD for 42 days.
  Interventions: Drug: Placebo for ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Capsule; oral
  Arms: Part A, ABBV-932; Part B, ABBV-932; Part C, ABBV-932; Part D, ABBV-932
Drug: Placebo for ABBV-932 — Capsule; oral
  Arms: Part A, Placebo for ABBV-932; Part B, Placebo for ABBV-932; Part C, Placebo for ABBV-932; Part D, Placebo for ABBV-932

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, safety, and tolerability following multiple ascending oral doses of ABBV-932 or placebo in healthy adult participants, participants with Generalized Anxiety Disorder (GAD), and participants with bipolar disorder (BPD).

ELIGIBILITY:
Inclusion Criteria:

* For healthy volunteer cohort:

  -- Body mass index (BMI) is >= 18.0 to <= 32.0 kg/m2 after rounding to the tenths decimal.
* For participants with generalized anxiety disorder (GAD) or bipolar disorder (BPD)

  * Participants with GAD or BPD (as confirmed by MINI) meet participant psychiatric history criteria described in the protocol.

Exclusion Criteria:

- History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 28
  Cmax will be assessed.
Time to Cmax (Tmax) | Up to Day 28
  Tmax will be assessed.
Plasma Concentrations at Pre-dose or at the End of a Dosing Interval (Ctrough) | Up to Day 28
  Ctrough will be assessed.
Area under the Plasma Concentration-time Curve from Time Zero to the End of the Dosing Interval (AUCtau) | Up to Day 28
  AUCtau will be assessed.
Number of Participants with Adverse Events (AEs) | Baseline to Day 129
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Collaborative Neuroscience Research CNS /ID# 260270, Los Alamitos, California
  - Acpru /Id# 255945, Grayslake, Illinois
  - Hassman Research Institute Marlton Site /ID# 260271, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-893